CLINICAL TRIAL: NCT01573000
Title: Phase II a Randomized Study of Iodine-131 Anti-b1 Antibody Versus Anti-b1 Antibody in Chemotherapy-relapsed/Refractory Low-grade or Transformed Low-grade Non-Hodgkin's Lymphoma (NHL)
Brief Title: A Randomized Study of Iodine-131 Anti-b1 Antibody Versus Anti-b1 Antibody in Chemotherapy-relapsed/Refractory Low-grade or Transformed Low-grade Non-Hodgkin's Lymphoma (NHL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 104515
Record Dates: First submitted 2012-03-08; First posted 2012-04-06 (Estimated); Results first posted 2012-10-05 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2016-11

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: Bexxar; Non-Hodgkin's Lymphoma; Tositumomab; Anti-B1 Antibody; Radioimmunotherapy; Iodine I-131; Iodine-131
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Open-label, two-arm, Arm A and Arm B Crossover (Experimental): Arm A Dosimetric Dose: 450 mg of TST infused over 70 minutes (inclusive of a 10-minute flush) immediately followed by 5 milliCurie (mCi) (35 mg) of I-131 TST infused over 30 minutes (inclusive of a 10-minute flush).• Therapeutic Dose: Seven to 14 days after the dosimetric dose, 450 mg of TST infused over 70 minutes (inclusive of a 10-minute flush) immediately followed by a subject-specific mCi activity (35 mg) of I-131 TST to deliver the desired total body dose (TBD) infused over 30 minutes (inclusive of a 10-minute flush). The desired TBD was 65 cGy for subjects with a baseline platelet count of 100,001-149,999 cells/mm3 and 75 cGy for subjects with a baseline platelet count ≥150,000 cells/mm3. Obese subjects (subjects weighing more than 137% of their calculated lean body weight) were dosed based upon 137% of their calculated lean body mass
  Interventions: Biological: Iodine-131 Anti-B1 Antibody Versus Anti-B1 Antibody in Chemotherapy-Relapsed/Refractory Low-Grade or Transformed Low-Grade Non-Hodgkin's Lymphoma (NHL)
- Arm B Crossover (Experimental): Arm B Dosimetric Dose: 450 mg of TST infused over 70 minutes (inclusive of a 10-minute flush) immediately followed by 35 mg of TST infused over 30 minutes (inclusive of a 10-minute flush).Therapeutic Dose: Seven to 14 days after the dosimetric dose, 450 mg of TST infused over 70 minutes (inclusive of a 10-minute flush) immediately followed by 35 mg of TST infused over 30 minutes (inclusive of a 10-minute flush). Subjects randomized to Arm B were allowed to cross-over and receive TST/ I-131 TST once their disease had progressed.
  Interventions: Biological: Iodine-131 Anti-B1 Antibody Versus Anti-B1 Antibody in Chemotherapy-Relapsed/Refractory Low-Grade or Transformed Low-Grade Non-Hodgkin's Lymphoma (NHL)

INTERVENTIONS:
Biological: Iodine-131 Anti-B1 Antibody Versus Anti-B1 Antibody in Chemotherapy-Relapsed/Refractory Low-Grade or Transformed Low-Grade Non-Hodgkin's Lymphoma (NHL) — Subjects will be randomized to receive tositumomab and iodine-131 tositumomab (Arm A) or unlabeled tositumomab (Arm B). Subjects randomized to receive unlabeled tositumomab may crossover and receive radiolabeled Iodine-131 tositumomab following progression of their lymphoma. Response in both arms will be assessed at 7 weeks, 13 weeks, and then at 3-monthly intervals for up to 2 years.

SUMMARY:
Subjects were randomized to receive either tositumomab (Anti-B1 Antibody) and iodine I 131 tositumomab (Arm A) or unlabeled tositumomab (Arm B). Subjects randomized to Arm B were allowed to cross over and receive I 131 tositumomab once their disease had progressed as long as they still fulfilled the protocol entry criteria (except for exclusion criterion 12, prior monoclonal antibody therapy) and were human anti-murine antibody (HAMA) negative. Study endpoint assessments of response were conducted by a Masked Independent Randomized Radiographic and Oncologic Review (MIRROR) panel and the Study Investigators' assessments of safety and survival. Subjects who completed at least two years of follow-up in Protocol BEX104515 (formerly Corixa Protocol RIT-II-002) were enrolled in long term follow-up Protocol BEX104526 (formerly Corixa Protocol CCBX001-051), an administrative protocol, for continued radiographic response evaluations and safety evaluations every 6 months for years 3 through 5 post-treatment and annually for years 6 through 10 post-treatment. Subjects in BEX104526 were assessed for survival, disease status, subsequent therapy for NHL, and long-term safety, including the use of thyroid medication, development of hypothyroidism, human anti murine antibody (HAMA), myelodysplastic syndrome, acute myelogenous leukemia, and all other secondary malignancies. Additionally, subjects were followed for the development of any adverse event(s) deemed by the Principal Investigator as being possibly or probably related to a subject's previous treatment with Iodine I-131 tositumomab. Laboratory evaluations consisting of a thyroid stimulating hormone level and a complete blood cell count, with a differential and platelet count, were obtained annually through year 10 post-treatment.

Dosimetric Dose: Subjects received 450 mg of tositumomab IV followed by 5.0 mCi of Iodine I-131 and 35 mg of tositumomab. Following the dosimetric dose, whole body dosimetry was performed on each subject using a total body gamma camera. Whole body anterior and posterior whole body images were obtained at the following timepoints.

1. Within one hour of infusion of the dosimetric dose and prior to urination
2. 2-4 days after infusion of the dosimetric dose, following urination
3. 6-7 days after infusion of the dosimetric dose, following urination Therapeutic Dose: The total body residence time, derived from total body gamma camera counts obtained at the 3 time points, was used to calculate the iodine-131 activity (mCi) to be administered to deliver the therapeutic total body irradiation dose of 65 or 75 cGy. The therapeutic step was administered 7-14 days after the dosimetric step and consisted of tositumomab 450 mg followed by an activity (mCi) of iodine-131 calculated to deliver 75 cGy or 65 cGy of total body irradiation, depending on platelet count, and 35 mg of tositumomab.

For subjects with ≥150,000 platelets/mm3, the recommended dose was the activity of iodine-131 calculated to deliver 75 cGy of total body irradiation; for subjects with NCI Grade 1 thrombocytopenia (platelet counts ≥100,000 but <150,000 platelets/mm3), the recommended dose was the activity of iodine-131 calculated to deliver 65 cGy of total body irradiation.

DETAILED DESCRIPTION:
This is a Phase II randomized, controlled, two-arm, open-label, multicenter study comparing the safety and efficacy of tositumomab and iodine I 131 tositumomab to tositumomab for the treatment of chemotherapy-relapsed or refractory low-grade or transformed low-grade B-cell NHL.

Treatment Arm A: Subject will undergo 2 phases of study. In the first phase, termed "dosimetric dose", subjects will receive tositumomab (450 mg) followed by tositumomab (35 mg) that has been trace labeled with 5mCi) Iodine-131 tositumomab. Whole body gamma camera scans will be obtained on day 0, day 2, 3, or 4, and day 6 or 7 following the dosimetric dose. Using the dosimetric data from three imaging time points, a subject-specific dose of iodine I 131 tositumomab to deliver the desired total body dose of radiotherapy will be calculated. In the second phase of the study, termed "therapeutic dose", subjects will receive unlabeled tositumomab (450mg) followed by iodine tositumomab (35mg) labeled with the subject-specific dose of iodine I-131 to deliver a whole body dose of 75 cGy to subjects. Subjects with platelet counts of 100,001 - 149,999 cells/mm3, will receive 65 cGy and subjects who are obese will be doses based on 137% of their lean body mass. Subjects will be treated with either saturated solution potassium iodide (SSKI), Lugol's solution, or potassium iodide tablets starting at least 24 hours prior to the first infusion of the Iodine-131 tositumomab (i.e., the dosimetric dose) and continuing for 14 days following the last infusion of radiolabeled tositumomab (i.e., the therapeutic dose).

Treatment Arm B: Subjects will receive the same amount of unlabeled tositumomab (450 + 35 mg) administered over the same time-frame as Arm A on the study Days 0 and 7 (the day 7 dose may be delayed but no longer than 14 days after the first dose).

Crossover treatment Arm B: Subjects in Arm B may crossover and receive Iodine-131 tositumomab following progression of their lymphoma if they still fulfill the protocol inclusion exclusion criteria (except exclusion criteria#12) and are HAMA-negative.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed low-grade or transformed NHL with evaluable, measurable disease
* Tumor had to express CD20 antigen
* One to three prior chemotherapy regimens
* Karnofsky performance score ≥60% and anticipated survival ≥3 months
* Absolute neutrophil count (ANC) >1500/mm3 and platelet count >100,000/mm3
* Adequate renal and hepatic function
* 18 years of age or older.
* Written informed consent and sign an IRB-approved Informed consent from prior to study entry.

Exclusion Criteria:

* More than an average of 25% of the intratrabecular marrow space involved by lymphoma in bone marrow biopsy specimens as assessed microscopically within 42 days of study entry. Bilateral posterior iliac crest core biopsies are required if the percentage of intratrabecular space involved exceeds 10% on a unilateral biopsy. The mean of bilateral biopsies must be no more than 25%.
* Received cytotoxic chemotherapy, radiation therapy, immunosuppressants, or cytokine treatment within FOUR weeks prior to study entry (6 weeks of nitrosourea compounds) or who exhibit persistent clinical evidence of toxicity. The use of steroids must be discontinued at least 1 week prior to study entry.
* Have undergone prior stem cell transplant.
* Active obstructive hydronephrosis.
* Evidence of active infection requiring intravenous antibiotics at the time of study entry.
* New York Heart Association class III or IV heart disease or other serious illness that would preclude evaluation.
* Prior malignancy other than lymphoma, except for adequately-treated skin cancer, in situ cervical cancer, or other cancer for which subject has been disease-free for 5 years.
* Known HIV infection.
* Known brain or leptomeningeal metastases.
* Pregnant or nursing. Subjects of childbearing potential must undergo pregnancy test within 7 days of study entry and antibody is not to be administered until a negative result is obtained. For those subjects in Arm B, the pregnancy test must be repeated within 7 days of crossover. Male and female must agree to use effective contraception for 6 months following the therapeutic dose, as applicable.
* Previous allergic reactions to iodine. This does not include reactions to intravenous iodine-containing contrast materials.
* Previously given any monoclonal or polyclonal antibodies of any non-human species for either diagnostic or therapeutic purpose. This includes engineered chimeric and humanized antibodies.
* Previously received radioimmunotherapy .
* Progressive disease within one year of irradiation arising in a field that has been previously irradiated with >3500 cGy.
* de novo intermediate or high-grade lymphoma.
* Received >3 chemotherapy regimens (different or identical agents).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 1998-09; Primary Completion 2001-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Result] Knox SJ, Goris ML, Davis TA, Trisler KD, Saal J, Levy R. Randomized controlled study of Iodine-131 Anti-B1 Antibody vs. unlabeled-Anti-B1 Antibody in subjects with chemotherapy refractory low-grade non-Hodgkin's Lymphoma [abstract]. Int J Radiat Oncol Biol Phys 1997;39(Suppl):326.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 104515 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 104515 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 104515 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 104515 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 104515 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 104515 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 104515 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants (par.) received radioimmunotherapy of tositumomab (TST)/Iodine I 131 TST (Arm A) or unlabeled TST (Arm B) in 2 phases: dosimetric and therapeutic dose. Arm B par. were allowed to crossover and receive I 131 TST, if disease progressed. After TST treatment, par. could have entered a Long-Term Follow-Up study (BEX104526; NCT00240591).
Groups:
- TST and Iodine I 131 TST: Participants received a dosimetric dose (DD) consisting of 450 milligrams (mg) of tositumomab (TST) intravenously (IV) followed by 5.0 millicurie (mCi) of Iodine I 131 and 35 mg of TST IV. The therapeutic dose (TD) consisting of 450 mg of TST IV, followed by a participant-specific dose of I 131 (75 centigray [cGy] or 65 cGy) and 35 mg of TST IV, was administered 7-14 days after the DD. Participants who had completed at least 2 years of follow-up after administration of TST/I 131 TST during the TD phase and had signed the informed consent to participate in the Long-Term Follow-Up (LTFU) study (BEX104526) were followed for up to 10 years. Participants did not receive any study medication during the LTFU study.
- Unlabeled TST: Participants received a DD consisting of 450 mg and 35 mg of unlabelled TST IV. The TD consisting of 450 mg and 35 mg of TST IV was administered 7-14 days after the DD. Participants randomized to receive 450 mg and 35 mg of unlabelled TST IV during the DD and TD phase were allowed to crossover and receive I 131 TST using the same regimen used in the TST and Iodine I 131 TST treatment arm once their disease had progressed as long as they still fulfilled the protocol entry criteria. Participants who had completed at least 2 years of follow-up after administration of TST during the TD phase and had signed the informed consent to participate in the LTFU study (BEX104526) were followed for up to 10 years. Participants did not receive any study medication during the LTFU study.
Period: Dosimetric and Therapeutic Treatment
Arm/Group | TST and Iodine I 131 TST | Unlabeled TST
Started | 42 | 36
Completed | 7 (These participants completed 2 years of follow up and enrolled in BEX104526.) | 1 (These participants completed 2 years of follow up and enrolled in BEX104526.)
Not Completed | 35 | 35
Not completed — Lack of Efficacy | 27 | 32
Not completed — Lost to Follow-up | 4 | 2
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Received Other Treatment | 2 | 0
Period: Crossover Phase
Arm/Group | TST and Iodine I 131 TST | Unlabeled TST
Started | 0 | 19 (19 of 36 par. randomized to receive Unlabeled TST crossed over to receive TST and Iodine I 131 TST.)
Completed | 0 | 1 (This participant completed 2 years of follow up and enrolled in BEX104526.)
Not Completed | 0 | 18
Not completed — Lack of Efficacy | 0 | 13
Not completed — Lost to Follow-up | 0 | 2
Not completed — Death | 0 | 3
Period: Long-Term Follow-Up
Arm/Group | TST and Iodine I 131 TST | Unlabeled TST
Started | 14 (14 of the 35 participants withdrawing from Study BEX104515 enrolled in long-term follow-up study.) | 5 (5 of the 35 participants withdrawing from Study BEX104515 enrolled in long-term follow-up study.)
Completed | 11 | 4 (One participant who received crossover treatment was lost to follow up.)
Not Completed | 3 | 1
Not completed — Death | 3 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TST and Iodine I 131 TST | Unlabeled TST | Total
Number analyzed (Participants) | 42 | 36 | 78
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.3 (11.6) | 55.4 (12.8) | 55.8 (12.1)
Sex/Gender, Customized [Number; unit: Participants]
  Female | 19 | 18 | 37
  Male | 23 | 18 | 41
Race/Ethnicity, Customized [Number; unit: participants]
  White | 39 | 33 | 72
  Hispanic | 1 | 1 | 2
  Asian | 0 | 1 | 1
  Black | 1 | 1 | 2
  Other/Unknown | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants (Par.) With Confirmed Response as Assessed by the Investigator
Description: Responses had to be confirmed by 2 separate evaluations occurring >=4 weeks apart. Par. with confirmed response include those with Complete Response (CR: complete resolution of all disease-related radiological abnormalities and the disappearance of all signs and symptoms related to the disease), Clinical Complete Response (CCR: complete resolution of all disease-related symptoms; residual foci, thought to be residual scar tissue, are present), or Partial Response (PR: >=50% reduction in the sum of the products of the longest perpendicular diameters of all measurable lesions; no new lesions).
Time Frame: Participants were evaluated for up to two years in Study BEX104515 and for up to 11.9 years in Study BEX104526.
Population: Intent-to-Treat (ITT) Exposed Population: all participants who were enrolled into the study and received at least one dose of study drug. Only those participants evaluable for confirmed response were analyzed.
Measure: Number; unit: participants
Groups:
- Unlabeled TST: Participants received a DD consisting of 450 mg and 35 mg of unlabelled TST IV. The TD consisting of 450 mg and 35 mg of TST IV was administered 7-14 days after the DD. Participants who had completed at least 2 years of follow-up after administration of TST during the TD phase and had signed the informed consent to participate in the LTFU study (BEX104526) were followed for up to 10 years. Participants did not receive any study medication during the LTFU study.
Arm/Group | TST and Iodine I 131 TST | Unlabeled TST
Number analyzed (Participants) | 36 | 27
participants | 21 | 8
Statistical Analysis 1: Comparison: TST and Iodine I 131 TST; Test type: Superiority or Other; percentage of participants = 50, 95% CI 2-sided [35 to 65] — The estimated value represents the percentage of participants with confirmed response (CR, CCR, PR). The number of participants evaluable for overall response (confirmed and unconfirmed; n=42) is used as the denominator
Statistical Analysis 2: Comparison: Unlabeled TST; Test type: Superiority or Other; percentage of participants = 22, 95% CI 2-sided [9 to 36] — The estimated value represents the percentage of participants with confirmed response (CR, CCR, PR). The number of participants evaluable for overall response (confirmed and unconfirmed; n=36) is used as the denominator

2. Primary Outcome: Number of Participants With Confirmed Response Before and After Crossover From Unlabeled TST to TST and Iodine I 131 TST as Assessed by the Investigator
Description: Participants receiving Unlabeled TST with progressive disease (defined as a >=25% increase from the nadir value of the sum of the products of the longest perpendicular diameters of all measureable lesions or the appearance of any new lesion. Individual lesions must be >2 centimeters [cm] in diameter by radiographic evaluation or >1 cm in diameter by physical examination.) were assessed separately before and after receiving the crossover treatment of I 131 TST for confirmed response, which included participants with CR, CCR, and PR.
Time Frame: Participants were evaluated for up to two years in Study BEX104515 and for up to 11.9 years in Study BEX104526.
Population: ITT-Exposed Population. All participants receiving Unlabeled TST who received the crossover treatment were analyzed.
Measure: Number; unit: participants
Groups:
- Unlabeled TST Crossover: Participants randomized to receive 450 mg and 35 mg of unlabelled TST IV during the DD and TD phase were allowed to crossover and receive I 131 TST using the same regimen used in the TST and Iodine I 131 TST treatment arm once their disease had progressed as long as they still fulfilled the protocol entry criteria. Participants who had completed at least 2 years of follow-up after administration of TST/I 131 TST during the TD phase and had signed the informed consent to participate in the LTFU study (BEX104526) were followed for up to 10 years. Participants did not receive any study medication during the LTFU study.
Arm/Group | Unlabeled TST | Unlabeled TST Crossover
Number analyzed (Participants) | 19 | 19
participants | 3 | 15
Statistical Analysis 1: Comparison: Unlabeled TST; Test type: Superiority or Other; percentage of participants = 16, 95% CI 2-sided [0 to 32] — The estimated value represents the percentage of participants with confirmed response (CR, CCR, PR) before Crossover
Statistical Analysis 2: Comparison: Unlabeled TST Crossover; Test type: Superiority or Other; percentage of participants = 79, 95% CI 2-sided [61 to 97] — The estimated value represents the percentage of participants with confirmed response (CR, CCR, PR) after Crossover

3. Primary Outcome: Number of Participants With Confirmed Complete Response (CR) as Assessed by the Investigator
Description: CR is defined as the complete resolution of all disease-related radiological abnormalities and the disappearance of all signs and symptoms related to the disease.
Time Frame: Participants were evaluated for up to two years in Study BEX104515 and for up to 11.9 years in Study BEX104526.
Population: ITT-Exposed Population. Only those participants evaluable for confirmed response were analyzed.
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST | Unlabeled TST
Number analyzed (Participants) | 36 | 27
participants | 11 | 3
Statistical Analysis 1: Comparison: TST and Iodine I 131 TST; Test type: Superiority or Other; percentage of participants = 26, 95% CI 2-sided [13 to 39] — The estimated value represents the percentage of participants with complete response. The number of participants evaluable for overall response (confirmed and unconfirmed; n=42) is used as the denominator
Statistical Analysis 2: Comparison: Unlabeled TST; Test type: Superiority or Other; percentage of participants = 8, 95% CI 2-sided [0 to 17] — The estimated value represents the percentage of participants with complete response. The number of participants evaluable for overall response (confirmed and unconfirmed; n=36) is used as the denominator

4. Primary Outcome: Number of Participants (Par.) With a Confirmed Complete Response as Assessed by the Masked Independent Randomized Radiology and Oncology Review (MIRROR) Panel
Description: as for outcome 1
Time Frame: The MIRROR panel reviewed responses of participants from 17 July 1998 to 17 January 2001
Population: ITT-Exposed Population. Only those participants evaluable for confirmed response were analyzed.
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST | Unlabeled TST
Number analyzed (Participants) | 42 | 36
participants | 14 | 3
Statistical Analysis 1: Comparison: TST and Iodine I 131 TST vs Unlabeled TST; Test type: Superiority or Other; p = 0.012, Fisher Exact

5. Primary Outcome: Number of Participants With Confirmed Complete Response (CR) Before and After Crossover From Unlabeled TST to TST and Iodine I 131 TST as Assessed by the Investigator
Description: Participants receiving Unlabeled TST with progressive disease were assessed separately before and after receiving the crossover treatment of I 131 TST for CR. CR is defined as the complete resolution of all disease-related radiological abnormalities and the disappearance of all signs and symptoms related to the disease.
Time Frame: Participants were evaluated for up to two years in Study BEX104515 and for up to 11.9 years in Study BEX104526.
Population: ITT-Exposed Population. All participants receiving Unlabeled TST who received the crossover treatment were analyzed.
Measure: Number; unit: participants
Arm/Group | Unlabeled TST | Unlabeled TST Crossover
Number analyzed (Participants) | 19 | 19
participants | 0 | 8
Statistical Analysis 1: Comparison: Unlabeled TST; Test type: Superiority or Other; percentage of participants = 0, 95% CI 2-sided [0 to 0] — The estimated value represents the percentage of participants with confirmed complete response before Crossover
Statistical Analysis 2: Comparison: Unlabeled TST Crossover; Test type: Superiority or Other; percentage of participants = 42, 95% CI 2-sided [20 to 64] — The estimated value represents the percentage of participants with confirmed complete response after Crossover

6. Primary Outcome: Number of Participants With Confirmed Clinical Complete Response (CCR) as Assessed by the Investigator
Description: CCR is defined as the complete resolution of all disease-related symptoms; residual foci, thought to be residual scar tissue, are present. Generally, an unchanging lesion =<2 cm in diameter by radiographic evaluation or =<1 cm in diameter by physical examination can be considered scar tissue.
Time Frame: Participants were evaluated for up to two years in Study BEX104515 and for up to 11.9 years in Study BEX104526.
Population: ITT-Exposed Population. Only those participants evaluable for confirmed response were analyzed.
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST | Unlabeled TST
Number analyzed (Participants) | 36 | 27
participants | 1 | 1
Statistical Analysis 1: Comparison: TST and Iodine I 131 TST; Test type: Superiority or Other; percentage of participants = 2, 95% CI 2-sided [0 to 7] — The estimated value represents the percentage of participants with confirmed CCR. The number of participants evaluable for overall response (confirmed and unconfirmed; n=42) is used as the denominator
Statistical Analysis 2: Comparison: Unlabeled TST; Test type: Superiority or Other; percentage of participants = 3, 95% CI 2-sided [0 to 8] — The estimated value represents the percentage of participants with confirmed CCR. The number of participants evaluable for overall response (confirmed and unconfirmed; n=36) is used as the denominator

7. Primary Outcome: Number of Participants With Confirmed Clinical Complete Response (CCR) Before and After Crossover From Unlabeled TST to TST and Iodine I 131 TST as Assessed by the Investigator
Description: Participants receiving Unlabeled TST with progressive disease were assessed separately before and after receiving the crossover treatment of I 131 TST for CCR. CCR is defined as the complete resolution of all disease-related symptoms; residual foci, thought to be residual scar tissue, are present. Generally, an unchanging lesion =<2 cm in diameter by radiographic evaluation or =<1 cm in diameter by physical examination can be considered scar tissue.
Time Frame: Participants were evaluated for up to two years in Study BEX104515 and for up to 11.9 years in Study BEX104526.
Population: ITT-Exposed Population. All participants receiving Unlabeled TST who received the crossover treatment were analyzed.
Measure: Number; unit: participants
Arm/Group | Unlabeled TST | Unlabeled TST Crossover
Number analyzed (Participants) | 19 | 19
participants | 0 | 1
Statistical Analysis 1: Comparison: Unlabeled TST; Test type: Superiority or Other; percentage of participants = 0, 95% CI 2-sided [0 to 0] — The estimated value represents the percentage of participants with confirmed CCR before Crossover
Statistical Analysis 2: Comparison: Unlabeled TST Crossover; Test type: Superiority or Other; percentage of participants = 5, 95% CI 2-sided [0 to 15] — The estimated value represents the percentage of participants with confirmed CCR after Crossover

8. Primary Outcome: Number of Participants With Confirmed Complete Response Plus Clinical Complete Response (CR + CCR) as Assessed by the Investigator
Description: CCR is defined as the complete resolution of all disease-related symptoms; residual foci, thought to be residual scar tissue, are present. Generally, an unchanging lesion =<2 cm in diameter by radiographic evaluation or =<1 cm in diameter by physical examination can be considered scar tissue. The extent of disease must be unchanged or decreased upon follow-up evaluations. If the extent of disease was unchanged or if further decreases occurred for 6 months or longer, the participant was reclassified as having a CR.
Time Frame: Participants were evaluated for up to two years in Study BEX104515 and for up to 11.9 years in Study BEX104526.
Population: ITT-Exposed Population. Only those participants evaluable for confirmed response were analyzed.
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST | Unlabeled TST
Number analyzed (Participants) | 36 | 27
participants | 13 | 4
Statistical Analysis 1: Comparison: TST and Iodine I 131 TST; Test type: Superiority or Other; percentage of participants = 31, 95% CI 2-sided [17 to 45] — The estimated value represents the percentage of participants with confirmed CR and CCR. The number of participants evaluable for overall response (confirmed and unconfirmed; n=42) is used as the denominator
Statistical Analysis 2: Comparison: Unlabeled TST; Test type: Superiority or Other; percentage of participants = 11, 95% CI 2-sided [1 to 21] — The estimated value represents the percentage of participants with confirmed CR and CCR. The number of participants evaluable for overall response (confirmed and unconfirmed; n=36) is used as the denominator

9. Primary Outcome: Number of Participants With Confirmed Complete Response Plus Clinical Complete Response (CR + CCR) Before and After Crossover From Unlabeled TST to TST and Iodine I 131 TST as Assessed by the Investigator
Description: Participants receiving Unlabeled TST with progressive disease were assessed separately before and after receiving the crossover treatment of I 131 TST for CR + CCR.
Time Frame: Participants were evaluated for up to two years in Study BEX104515 and for up to 11.9 years in Study BEX104526.
Population: ITT-Exposed Population. All participants receiving Unlabeled TST who received the crossover treatment were analyzed.
Measure: Number; unit: participants
Arm/Group | Unlabeled TST | Unlabeled TST Crossover
Number analyzed (Participants) | 19 | 19
participants | 0 | 9
Statistical Analysis 1: Comparison: Unlabeled TST; Test type: Superiority or Other; percentage of participants = 0, 95% CI 2-sided [0 to 0] — The estimated value represents the percentage of participants with confirmed CR and CCR before Crossover
Statistical Analysis 2: Comparison: Unlabeled TST Crossover; Test type: Superiority or Other; percentage of participants = 47, 95% CI 2-sided [25 to 70] — The estimated value represents the percentage of participants with confirmed CR and CCR after Crossover

10. Primary Outcome: Number of Participants With Confirmed Partial Response (PR) as Assessed by the Investigator
Description: Confirmed PR is defined as a >=50% reduction in the sum of the products of the longest perpendicular diameters of all measurable lesions, with no new lesions.
Time Frame: Participants were evaluated for up to two years in Study BEX104515 and for up to 11.9 years in Study BEX104526.
Population: ITT-Exposed Population. Only those participants evaluable for confirmed response were analyzed.
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST | Unlabeled TST
Number analyzed (Participants) | 36 | 27
participants | 7 | 4
Statistical Analysis 1: Comparison: TST and Iodine I 131 TST; Test type: Superiority or Other; percentage of participants = 17, 95% CI 2-sided [5 to 28] — The estimated value represents the percentage of participants with confirmed PR. The number of participants evaluable for overall response (confirmed and unconfirmed; n=42) is used as the denominator
Statistical Analysis 2: Comparison: Unlabeled TST; Test type: Superiority or Other; percentage of participants = 11, 95% CI 2-sided [1 to 21] — The estimated value represents the percentage of participants with confirmed PR. The number of participants evaluable for overall response (confirmed and unconfirmed; n=36) is used as the denominator

11. Secondary Outcome: Number of Participants (Par.) With a Confirmed Response (CR, CCR, or PR) as Assessed by the MIRROR Panel
Description: as for outcome 1
Time Frame: The MIRROR panel reviewed responses of participants from 17 July 1998 to 17 January 2001
Population: ITT-Exposed Population. Only those participants evaluable for confirmed response were analyzed.
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST | Unlabeled TST
Number analyzed (Participants) | 42 | 36
participants | 23 | 6
Statistical Analysis 1: Comparison: TST and Iodine I 131 TST vs Unlabeled TST; Test type: Superiority or Other; p = 0.001, Fisher Exact

12. Secondary Outcome: Duration of Response for All Confirmed Responders, Confirmed Complete Responders, and Confirmed Partial Responders
Description: For all participants with CR, CCR, or PR, duration of response was defined as the time from first documented response to first documented progression. All confirmed responders included participants with CR, CCR, and PR, whereas confirmed complete responders included participants with CR and CCR.
Time Frame: Participants were evaluated for up to two years in Study BEX104515 and for up to 11.9 years in Study BEX104526.
Population: ITT-Exposed Population. Only those participants evaluable for CR, CCR, or PR were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TST and Iodine I 131 TST | Unlabeled TST
Number analyzed (Participants) | 21 | 8
months
  All Confirmed Responders, n=21, 8 | 42.0 [9.0 to 116.8] | 18.5 [4.8 to NA] — The upper limit of the 95% confidence interval (CI) was not able to be determined (not reached) because there were not enough events to be able to calculate the upper limit of the 95% CI.
  Confirmed Complete Responders, n=13, 4 | 116.8 [58.5 to NA] — The upper limit of the 95% confidence interval (CI) was not able to be determined (not reached) because there were not enough events to be able to calculate the upper limit of the 95% CI. | NA [NA to NA] — The median (and 95% CI) from a Kaplan Meier survival curve cannot be determined if more than half the participants are censored (i.e., still alive or in continued response) when the study ends.
  Confirmed PR, n=7, 4 | 4.6 [3.0 to 9.0] | 6.2 [3.7 to 8.9]

13. Secondary Outcome: MIRROR Panel Assessments of Duration of Complete Response (Time From the First Documented Response to the First Documented Progression)
Description: as for outcome 1
Time Frame: The MIRROR panel reviewed responses of participants from 17 July 1998 to 17 January 2001
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TST and Iodine I 131 TST | Unlabeled TST
Number analyzed (Participants) | 42 | 36
months | NA [NA to NA] — The median (and 95% CI) from a Kaplan Meier survival curve cannot be determined if more than half the participants are censored (i.e., still alive or in continued response) when the study ends. | NA [28.1 to NA] — The median (and 95% CI) from a Kaplan Meier survival curve cannot be determined if more than half the participants are censored (i.e., still alive or in continued response) when the study ends.
Statistical Analysis 1: Comparison: TST and Iodine I 131 TST vs Unlabeled TST; Test type: Superiority or Other; p = 0.495, Log Rank

14. Secondary Outcome: MIRROR Panel Assessments of Duration of Confirmed Response (Time From the First Documented Response to the First Documented Progression)
Description: as for outcome 1
Time Frame: The MIRROR panel reviewed responses of participants from 17 July 1998 to 17 January 2001
Population: ITT-Exposed Population. Only those participants evaluable for confirmed response were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TST and Iodine I 131 TST | Unlabeled TST
Number analyzed (Participants) | 42 | 36
months | NA [7.4 to NA] — The median (and 95% CI) from a Kaplan Meier survival curve cannot be determined if more than half the participants are censored (i.e., still alive or in continued response) when the study ends. | 18 [7.6 to NA] — The upper limit of the 95% confidence interval (CI) was not able to be determined (not reached) because there were not enough events to be able to calculate the upper limit of the 95% CI.
Statistical Analysis 1: Comparison: TST and Iodine I 131 TST vs Unlabeled TST; Test type: Superiority or Other; p = 0.677, Log Rank

15. Secondary Outcome: Time to Progression of Disease or Death as Assessed by the Investigator
Description: Progression-free survival or time to progression is defined as the time from the dosimetric dose to the first documented occurrence of disease progression or death.
Time Frame: Participants were evaluated for up to two years in Study BEX104515 and for up to 11.9 years in Study BEX104526.
Population: ITT-Exposed Population. Participants who experienced progression or died (n=36, 33) and participants who were censored (n=6, 3) were analyzed. A censored value indicates that the participant did not have the event of interest.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TST and Iodine I 131 TST | Unlabeled TST
Number analyzed (Participants) | 42 | 36
months | 6.0 [3.3 to 11.1] | 3.8 [2.9 to 6.0]

16. Secondary Outcome: Time to Progression of Disease or Death in Participants Before and After Crossover From Unlabeled TST to TST and Iodine I 131 TST as Assessed by the Investigator
Description: as for outcome 15
Time Frame: Participants were evaluated for up to two years in Study BEX104515 and for up to 11.9 years in Study BEX104526.
Population: ITT-Exposed Population. All participants receiving Unlabeled TST who received the crossover treatment and those who progressed/died were analyzed. Participants who experienced progression or died (n=18, 17) and participants who were censored (n=1, 2) were analyzed. A censored value indicates that the participant did not have the event of interest.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Unlabeled TST | Unlabeled TST Crossover
Number analyzed (Participants) | 19 | 19
months | 3.1 [2.8 to 6.0] | 15.0 [6.4 to 25.6]

17. Secondary Outcome: MIRROR Panel Assessed Time to Response (Time From the Date of Enrollment to the First Documented Response (PR, CR, CCR)
Description: as for outcome 1
Time Frame: The MIRROR panel reviewed responses of participants from 17 July 1998 to 17 January 2001
Population: ITT-Exposed Population. Only those participants evaluable for confirmed response were analyzed.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | TST and Iodine I 131 TST | Unlabeled TST
Number analyzed (Participants) | 42 | 36
days | 49 [48 to 54] | 69 [50 to 90]
Statistical Analysis 1: Comparison: TST and Iodine I 131 TST vs Unlabeled TST; Test type: Superiority or Other; p = 0.119, Log Rank

18. Secondary Outcome: MIRROR Panel Assessed Progression-free Survival
Description: Time from the date of enrollment (the date of randomization) to the first documented progression or death.
Time Frame: The MIRROR panel reviewed responses of participants from 17 July 1998 to 17 January 2001
Population: ITT-Exposed Population. Only those participants evaluable for confirmed response were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TST and Iodine I 131 TST | Unlabeled TST
Number analyzed (Participants) | 42 | 36
months | 6.3 [4.9 to NA] — The upper limit of the 95% confidence interval (CI) was not able to be determined (not reached) because there were not enough events to be able to calculate the upper limit of the 95% CI. | 5.5 [2.9 to 6.0]
Statistical Analysis 1: Comparison: TST and Iodine I 131 TST vs Unlabeled TST; Test type: Superiority or Other; p = 0.016, Log Rank

19. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from the treatment start date to the date of death by any cause.
Time Frame: Participants were evaluated for up to two years in Study BEX104515 and for up to 11.9 years in Study BEX104526.
Population: ITT-Exposed Population. Only those participants who died during the study and during the follow-up period were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TST and Iodine I 131 TST | Unlabeled TST | Unlabeled TST Crossover
Number analyzed (Participants) | 25 | 10 | 13
months | 71.5 [25.3 to NA] — The upper limit of the 95% confidence interval (CI) was not able to be determined (not reached) because there were not enough events to be able to calculate the upper limit of the 95% CI. | 70.0 [30.9 to NA] — The upper limit of the 95% confidence interval (CI) was not able to be determined (not reached) because there were not have enough events to be able to calculate the upper limit of the 95% CI. | 51.4 [19.3 to 86.4]

20. Secondary Outcome: Number of Participants With the Indicated Drug-Related (DR) Adverse Events (AEs) Experienced by 3 or More Participants
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. Causality of AEs was determined by the investigators as "none," "remote," "possible," "probable," or "highly probable." AEs considered by the investigator as being at least remotely related to the study treatment were considered to be DR AEs. White blood cell (WBC) count and absolute neutrophil count (ANC) were measured as cells per millimeters cubed (mm^3); hemoglobin was measured in grams per deciliter (g/dL).
Time Frame: Participants were evaluated for up to two years in Study BEX104515 and for up to 11.9 years in Study BEX104526.
Population: ITT-Exposed Population. All participants with any drug-related adverse events were analyzed.
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST | Unlabeled TST | Unlabeled TST Crossover
Number analyzed (Participants) | 42 | 32 | 17
participants
  Fatigue | 12 | 11 | 6
  Pyrexia | 12 | 6 | 3
  Chills | 10 | 7 | 3
  Pain | 2 | 3 | 1
  Malaise | 3 | 0 | 1
  Asthenia | 2 | 1 | 0
  Chest discomfort | 2 | 1 | 0
  Feeling hot | 1 | 2 | 0
  Oedema peripheral | 1 | 2 | 0
  Influenza like illness | 1 | 1 | 1
  Nausea | 20 | 5 | 2
  Diarrhoea | 4 | 1 | 1
  Abdominal discomfort | 2 | 1 | 2
  Dyspepsia | 3 | 0 | 2
  Vomiting | 2 | 2 | 0
  Abdominal pain upper | 3 | 0 | 0
  Constipation | 3 | 0 | 0
  WBC <2000 cells/mm^3 | 18 | 4 | 11
  ANC <1000 cells/mm^3 | 14 | 4 | 11
  Platelates <50000 cells/mm^3 | 15 | 1 | 9
  Hemoglobin < 8.0 g/dL | 6 | 0 | 3
  Rash | 5 | 2 | 2
  Erythema | 3 | 2 | 0
  Pruritus | 1 | 3 | 2
  Hyperhidrosis | 3 | 1 | 1
  Urticaria | 1 | 3 | 0
  Night sweats | 2 | 0 | 1
  Cough | 3 | 1 | 4
  Throat irritation | 2 | 2 | 2
  Oropharyngeal pain | 4 | 0 | 1
  Nasal congestion | 1 | 2 | 2
  Dyspnoea | 2 | 0 | 1
  Sinus congestion | 1 | 1 | 1
  Arthralgia | 8 | 5 | 2
  Myalgia | 8 | 5 | 0
  Back pain | 2 | 2 | 1
  Neck pain | 2 | 0 | 1
  Upper respiratory tract infection | 3 | 2 | 1
  Pneumonia | 2 | 1 | 1
  Bronchitis | 1 | 1 | 1
  Sinusitis | 0 | 1 | 2
  Headache | 5 | 5 | 4
  Dizziness | 3 | 2 | 0
  Paraesthesia | 1 | 1 | 1
  Thrombocytopenia | 6 | 0 | 3
  Anaemia | 5 | 0 | 2
  Lymphadenopathy | 3 | 3 | 0
  Lymph node pain | 2 | 1 | 1
  Neutropenia | 2 | 0 | 1
  Pancytopenia | 1 | 0 | 2
  Myelodysplastic syndrome | 3 | 0 | 4
  Basal cell carcinoma | 1 | 1 | 1
  Body temperature increased | 3 | 1 | 0
  Weight decreased | 2 | 0 | 1
  Insomnia | 4 | 2 | 0
  Decreased appetite | 6 | 2 | 0
  Flushing | 2 | 1 | 0
  Hypothyroidism | 3 | 0 | 3
  Ear pruritus | 1 | 1 | 1

21. Secondary Outcome: Number of Participants With the Indicated Type of Infection
Description: An infection is the colonization of a host organism by a parasite species. Infecting parasites seek to use the host's resources to reproduce, often resulting in disease. Specimen samples of the body fluid are cultured for testing whether the infectious organism is present and grown in the culture media to assess the growth pattern of the organisms present in the specimen. The culture results could be positive or negative. The positive culture results indicate that the tested participant has the infection under investigation, in which case therapeutic treatment with anti-infective is required.
Time Frame: Participants were evaluated for up to two years in Study BEX104515 and for up to 11.9 years in Study BEX104526.
Population: ITT-Exposed Population
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST | Unlabeled TST | Unlabeled TST Crossover
Number analyzed (Participants) | 42 | 36 | 19
participants
  Any Infection; n=42, 36, 19 | 18 | 9 | 7
  No Infection; n=42, 36, 19 | 24 | 27 | 12
  Sepsis; n=18, 9, 7 | 2 | 0 | 0
  Pneumonia; n=18, 9, 7 | 2 | 2 | 0
  Endocarditis/pericarditis; n=18, 9, 7 | 0 | 1 | 0
  Peritonitis; n=18, 9, 7 | 0 | 0 | 0
  Other infections; n=18, 9, 7 | 17 | 8 | 7

22. Secondary Outcome: Number of Participants With an Infection for Which Anti-infectives Were Administered
Description: Anti-infectives are capable of acting against infection, by inhibiting the spread of an infectious agent or by killing the infectious agent outright. Anti-infective is a general term that encompasses antibacterials, antibiotics, antifungals, antiprotozoans, and antivirals.
Time Frame: Participants were evaluated for up to two years in Study BEX104515 and for up to 11.9 years in Study BEX104526.
Population: ITT-Exposed Population. Only those participants who had an infection during the study and during the follow-up period were analyzed.
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST | Unlabeled TST | Unlabeled TST Crossover
Number analyzed (Participants) | 18 | 9 | 7
participants
  Anti-infective Administered | 16 | 9 | 6
  Anti-infective Not Administered | 2 | 0 | 1

23. Secondary Outcome: Number of Participants With the Indicated Grade 3 or Grade 4 AEs Experienced by 3 or More Participants
Description: AEs were graded using the Common Toxicity Criteria from the Cancer Therapy Evaluation Program, Division of Cancer Therapy, National Cancer Institute. Grades: 0 = No adverse event or within normal limits; 1 = Mild adverse event; 2 = Moderate adverse event; 3 = Severe and undesirable adverse event; 4 = Life-threatening or disabling adverse event; 5 = Death related to adverse event.
Time Frame: Participants were evaluated for up to two years in Study BEX104515 and for up to 11.9 years in Study BEX104526.
Population: ITT-Exposed Population. All participants with any Grade 3 or Grade 4 AEs experienced by 3 or more participants were analyzed.
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST | Unlabeled TST | Unlabeled TST Crossover
Number analyzed (Participants) | 32 | 12 | 14
participants
  WBC <2000 cells/mm^3 | 18 | 4 | 11
  ANC <1000 cells/mm^3 | 14 | 4 | 11
  Platelets <50000 cells/mm^3 | 15 | 1 | 9
  Hemoglobin <8.0 g/dL | 6 | 0 | 3
  Myelodysplastic syndrome | 4 | 0 | 4
  Basal cell carcinoma | 1 | 1 | 1
  Thrombocytopenia | 5 | 0 | 2
  Anaemia | 2 | 0 | 1
  Neutropenia | 2 | 0 | 1
  Pancytopenia | 1 | 0 | 2
  Pneumonia | 1 | 2 | 1
  Dyspnoea | 2 | 1 | 0

24. Secondary Outcome: Number of Participants With the Indicated Grade 3 or Grade 4 Drug-related AEs Experienced by 3 or More Participants
Description: as for outcome 23
Time Frame: Participants were evaluated for up to two years in Study BEX104515 and for up to 11.9 years in Study BEX104526.
Population: ITT-Exposed Population. All participants with any Grade 3 or Grade 4 drug-related AEs experienced by 3 or more participants were analyzed.
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST | Unlabeled TST | Unlabeled TST Crossover
Number analyzed (Participants) | 30 | 11 | 14
participants
  WBC <2000 cells/mm^3 | 18 | 4 | 11
  ANC <1000 cells/mm^3 | 14 | 4 | 11
  Platelets <50000 cells/mm^3 | 15 | 1 | 9
  Hemoglobin <8.0 g/dL | 6 | 0 | 3
  Myelodysplastic Syndrome | 3 | 0 | 4
  Basal Cell Carcinoma | 1 | 1 | 1
  Thrombocytopenia | 5 | 0 | 2
  Anaemia | 2 | 0 | 1
  Neutropenia | 2 | 0 | 1
  Pancytopenia | 1 | 0 | 2
  Pneumonia | 1 | 1 | 1

25. Secondary Outcome: Number of Participants With the Indicated Primary Cause of Death
Description: Participants were categorized according to their primary cause of death. Deaths due to progressive disease or to another reason ("Other") were not captured as serious adverse events (SAEs) and are thus not included in the SAE module.
Time Frame: Participants were evaluated for up to two years in Study BEX104515 and for up to 11.9 years in Study BEX104526.
Population: ITT-Exposed Population. All participants who died by the completion of LTFU were analyzed.
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST | Unlabeled TST | Unlabeled TST Crossover
Number analyzed (Participants) | 25 | 10 | 13
participants
  Unknown | 1 | 1 | 1
  Progression of lymphoma | 17 | 6 | 9
  Other | 7 | 3 | 3

26. Secondary Outcome: Number of Participants With a Time to Death From the Last Dose of Study Drug Less Than or Equal to 30 Days or More Than 30 Days
Description: Time to death from the last dose of study drug is the time from the last dose of study drug administered to the date of death. Deaths due to progressive disease or to another reason ("Other") were not captured as serious adverse events (SAEs) and are thus not included in the SAE module.
Time Frame: Participants were evaluated for up to two years in Study BEX104515 and for up to 11.9 years in Study BEX104526.
Population: ITT-Exposed Population. All participants who died by the completion of LTFU were analyzed.
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST | Unlabeled TST | Unlabeled TST Crossover
Number analyzed (Participants) | 25 | 10 | 13
participants
  =<30 Days | 0 | 0 | 0
  >30 Days | 25 | 10 | 13

27. Secondary Outcome: Number of Participants With the Indicated Serious Adverse Events (SAE) Related to Study Drug
Description: An SAE is any event occurring at any dose that results in any of the following: death, a life-threatening adverse drug experience (ADE; at immediate risk of death from the experience as it occurred), inpatient hospitalization/prolongation of existing hospitalization, a persistent/significant disability/incapacity, or a congenital anomaly/birth defect. Medical events that may not result in death, be life-threatening, or require hospitalization may be considered to be a serious ADEs when based upon appropriate medical judgment. Relatedness was based on the investigator's medical judgement.
Time Frame: Participants were evaluated for up to two years in Study BEX104515 and for up to 11.9 years in Study BEX104526.
Population: ITT-Exposed Population. All participants who experienced any SAE were analyzed.
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST | Unlabeled TST | Unlabeled TST Crossover
Number analyzed (Participants) | 18 | 6 | 10
participants
  Myelodysplastic Syndrome | 3 | 0 | 4
  Basal cell carcinoma | 1 | 1 | 1
  Bacteraemia | 2 | 0 | 0
  Acute myeloid leukaemia | 2 | 0 | 0
  Pancytopenia | 1 | 0 | 1
  Pneumonia | 1 | 0 | 1
  Squamous cell carcinoma | 0 | 0 | 1
  Abdominal pain upper | 1 | 0 | 0
  Back pain | 1 | 0 | 0
  Burkitt's lymphoma | 1 | 0 | 0
  Cholecystitis acute | 1 | 0 | 0
  Constipation | 1 | 0 | 0
  Cystitis | 0 | 1 | 0
  Febrile neutropenia | 0 | 1 | 0
  Gastrointestinal haemorrhage | 1 | 0 | 0
  Hypothermia | 0 | 1 | 0
  Mental status changes | 0 | 1 | 0
  Myocardial infarction | 0 | 1 | 0
  Proteus infection | 1 | 0 | 0
  Pyrexia | 1 | 0 | 0
  Renal cancer | 1 | 0 | 0
  Retroperitoneal haemorrhage | 0 | 1 | 0
  Small intestinal obstruction | 1 | 0 | 0
  Spinal cord compression | 1 | 0 | 0
  Syncope | 0 | 1 | 0
  Bronchitis | 0 | 0 | 1
  Chronic myelomonocytic leukaemia | 0 | 0 | 1
  Haemoptysis | 0 | 0 | 1
  Squamous cell carcinoma of skin | 0 | 0 | 1
  Subdural haematoma | 0 | 0 | 1
  Thrombocytopenia | 0 | 0 | 1
  Ulcer | 0 | 0 | 1

28. Secondary Outcome: Number of Participants With the Indicated Fatal SAEs Related to Study Drug
Description: as for outcome 27
Time Frame: Participants were evaluated for up to two years in Study BEX104515 and for up to 11.9 years in Study BEX104526.
Population: ITT-Exposed Population. All participants who experienced any fatal SAE were analyzed.
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST | Unlabeled TST | Unlabeled TST Crossover
Number analyzed (Participants) | 5 | 3 | 6
participants
  Myelodysplastic syndrome | 2 | 0 | 3
  Acute myeloid leukemia | 1 | 0 | 0
  Chronic myelomonocytic leukaemia | 0 | 0 | 1
  Thrombocytopenia | 0 | 0 | 1

29. Secondary Outcome: Time to Nadir and Time to Recovery to Baseline in Hematologic Laboratory Evaluations
Description: Nadir is defined as the lowest laboratory value recorded following the administration of the study medication. Time to recovery to baseline in hematologic laboratory evaluations is the time required for recovery from nadir values to baseline values. Hematologic laboratory evaluations included ANC, hemoglobin (Hb), platelets (Plt), and WBC count.
Time Frame: Participants were evaluated for up to two years in Study BEX104515 and for up to 11.9 years in Study BEX104526.
Population: ITT-Exposed Population. All participants with hematological toxicity were evaluated. The numbers analyzed in the category titles reflect the number of participants with the event of interest plus the number of participants who were censored. A censored value indicates that the participant did not have the event of interest.
Measure: Median (Full Range); unit: days
Arm/Group | TST and Iodine I 131 TST | Unlabeled TST | Unlabeled TST Crossover
Number analyzed (Participants) | 42 | 36 | 19
days
  Time to nadir ANC, n=42, 35, 19 | 48 [9 to 91] | 39 [8 to 91] | 44 [14 to 69]
  Time to nadir Hb, n=42, 36, 19 | 49 [9 to 112] | 43.5 [13 to 98] | 48 [14 to 115]
  Time to nadir Plt, n=42, 36, 19 | 36.5 [6 to 49] | 43.5 [7 to 112] | 36 [26 to 117]
  Time to nadir WBC count, n=42, 36, 19 | 46.5 [9 to 91] | 42.5 [8 to 91] | 43 [14 to 69]
  Time to recovery to baseline ANC, n=42, 35, 19 | 63 [56 to 75] | 41 [26 to 56] | 84 [63 to 97]
  Time to recovery to baseline Hb, n=42, 36, 19 | 69 [55 to 85] | 49 [33 to 58] | 97 [55 to 273]
  Time to recovery to baseline Plt, n=42, 36, 19 | 55 [49 to 61] | 44 [26 to 56] | 62.5 [49 to NA] — The upper limit of the 95% confidence interval (CI) was not able to be determined (not reached) because there were not enough events to be able to calculate the upper limit of the 95% CI.
  Time to recovery to baseline WBC, n=42, 36, 19 | 76 [65 to 105] | 54 [35 to 58] | 91 [75 to 168]

30. Secondary Outcome: Nadir Values for ANC, a Hematologic Parameter
Description: Nadir is defined as the lowest laboratory value recorded following the administration of study medication. ANC is a measure of the number of neutrophil granulocytes present in the blood. Neutrophils are a type of white blood cell that fights against infection.
Time Frame: Participants were evaluated for up to two years in Study BEX104515 and for up to 11.9 years in Study BEX104526.
Population: ITT-Exposed Population. All participants with hematological toxicity were evaluated.
Measure: Median (Full Range); unit: Cells/millimeters cubed (mm^3)
Arm/Group | TST and Iodine I 131 TST | Unlabeled TST | Unlabeled TST Crossover
Number analyzed (Participants) | 42 | 35 | 19
Cells/millimeters cubed (mm^3) | 1.3 [0 to 6] | 2.6 [0 to 5] | 0.8 [0 to 4]

31. Primary Outcome: Number of Participants With Confirmed Partial Response (PR) Before and After Crossover From Unlabeled TST to TST and Iodine I 131 TST as Assessed by the Investigator
Description: Participants receiving Unlabeled TST with progressive disease were assessed separately before and after receiving the crossover treatment of I 131 TST confirmed PR. Confirmed PR is defined as a >=50 percent reduction in the sum of the products of the longest perpendicular diameters of all measurable lesions, with no new lesions.
Time Frame: Participants were evaluated for up to two years in Study BEX104515 and for up to 11.9 years in Study BEX104526.
Population: ITT-Exposed Population. All participants receiving Unlabeled TST who received the crossover treatment were analyzed.
Measure: Number; unit: participants
Arm/Group | Unlabeled TST | Unlabeled TST Crossover
Number analyzed (Participants) | 19 | 19
participants | 3 | 6
Statistical Analysis 1: Comparison: Unlabeled TST; Test type: Superiority or Other; percentage of participants = 16, 95% CI 2-sided [0 to 32] — The estimated value represents the percentage of participants with confirmed PR before Crossover
Statistical Analysis 2: Comparison: Unlabeled TST Crossover; Test type: Superiority or Other; percentage of participants = 32, 95% CI 2-sided [11 to 52] — The estimated value represents the percentage of participants with confirmed PR after Crossover

32. Secondary Outcome: Nadir Values for Hemoglobin, a Hematologic Parameter
Description: Nadir is defined as the lowest laboratory value recorded following the administration of study medication. Hemoglobin is the iron-containing oxygen-transport metalloprotein in the red blood cells.
Time Frame: Participants were evaluated for up to two years in Study BEX104515 and for up to 11.9 years in Study BEX104526.
Population: ITT-Exposed Population
Measure: Median (Full Range); unit: Grams/dL
Arm/Group | TST and Iodine I 131 TST | Unlabeled TST | Unlabeled TST Crossover
Number analyzed (Participants) | 42 | 36 | 19
Grams/dL | 11 [6 to 14] | 12.5 [8 to 15] | 10.2 [7 to 14]

33. Secondary Outcome: Nadir Values for the Hematologic Parameters Platelets and WBC Count
Description: Nadir is defined as the lowest laboratory value recorded following the administration of study medication. Platelets and WBCs are types of blood cells.
Time Frame: Participants were evaluated for up to two years in Study BEX104515 and for up to 11.9 years in Study BEX104526.
Population: ITT-Exposed Population
Measure: Median (Full Range); unit: cells/microliter
Arm/Group | TST and Iodine I 131 TST | Unlabeled TST | Unlabeled TST Crossover
Number analyzed (Participants) | 42 | 36 | 19
cells/microliter
  Platelets (10000 cells/microliter) | 69 [5 to 261] | 162.5 [68 to 403] | 50 [12 to 138]
  WBC count (1000 cells/microliter) | 2.3 [1 to 7] | 4.4 [1 to 13] | 1.7 [1 to 5]

34. Secondary Outcome: Number of Participants With the Indicated Grade 3 or Grade 4 Hematologic Toxicities
Description: Adverse events were graded using the Common Toxicity Criteria from the Cancer Therapy Evaluation Program, Division of Cancer Therapy, National Cancer Institute. Grades: 0 = No adverse event or within normal limits; 1 = Mild adverse event; 2 = Moderate adverse event; 3 = Severe and undesirable adverse event; 4 = Life-threatening or disabling adverse event; 5 = Death related to adverse event.
Time Frame: Participants were evaluated for up to two years in Study BEX104515 and for up to 11.9 years in Study BEX104526.
Population: ITT-Exposed Population
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST | Unlabeled TST | Unlabeled TST Crossover
Number analyzed (Participants) | 42 | 36 | 19
participants
  ANC | 14 | 4 | 11
  Hemoglobin | 6 | 0 | 3
  Platelets | 15 | 1 | 9
  WBC count | 18 | 4 | 11

35. Secondary Outcome: Duration of the Indicated Grade 3 or Grade 4 Hematologic Toxicities
Description: as for outcome 34
Time Frame: Participants were evaluated for up to two years in Study BEX104515 and for up to 11.9 years in Study BEX104526.
Population: ITT-Exposed Population. All participants with Grade 3 or Grade 4 hematologic toxicities were analyzed. The "n" in the category titles reflects the number of participants with the indicated Grade 3 or Grade 4 hematologic toxicity.
Measure: Median (Full Range); unit: days
Arm/Group | TST and Iodine I 131 TST | Unlabeled TST | Unlabeled TST Crossover
Number analyzed (Participants) | 42 | 36 | 19
days
  ANC, n=14, 4, 11 | 15 [6 to 128] | 24 [2 to 36] | 16 [6 to 541]
  Hemoglobin, n=6, 0, 3 | 16 [8 to 71] | NA [NA to NA] — No participants had grade 3 or grade 4 hematologic toxicities in this arm. | 42 [18 to 98]
  Platelets, n=15, 1, 9 | 22 [7 to 314] | 411 [411 to 411] | 41 [8 to 195]
  WBC count, n=18, 4, 11 | 20 [6 to 326] | 22 [4 to 252] | 30 [14 to 503]

36. Secondary Outcome: Time to Human Anti-Murine Antibodies (HAMA) Positivity From the First Dosimetric Dose
Description: Tositumomab is a murine (mouse) antibody (immunoglobulin) of the IgG2a subclass. Participants in this study were evaluated to determine whether they developed an immune response to study treatment as evident by human anti-mouse antibodies (HAMA) after administration of tositumomab and iodine I 131 tositumomab. A positive HAMA value indicates that the participant developed human anti-mouse antibodies above the HAMA assay threshold, and a negative HAMA value indicates either the absence or below threshold level of human anti-mouse antibodies.
Time Frame: Participants were evaluated for up to two years in Study BEX104515 and for up to 11.9 years in Study BEX104526.
Population: ITT-Exposed Population. Participants who converted from being negative for HAMA at Baseline to being positive for HAMA following treatment were evaluated.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | TST and Iodine I 131 TST | Unlabeled TST | Unlabeled TST Crossover
Number analyzed (Participants) | 13 | 10 | 0
days | 163 (108.4) | 62.6 (49) |

ADVERSE EVENTS:
Time Frame: Participants were evaluated for up to two years in Study BEX104515 and for up to 11.9 years in Study BEX104526.
Description: Serious adverse events are reported regardless of causality. Deaths due to progressive disease or to another reason ("Other") were not captured as serious adverse events (SAEs) and are thus not included in the SAE module.
Arm/Group | TST and Iodine I 131 TST | Unlabeled TST | Unlabeled TST Crossover
Serious Adverse Events (participants affected / at risk) | 18/42 | 6/36 | 10/19
Other Adverse Events (participants affected / at risk) | 42/42 | 33/36 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TST and Iodine I 131 TST (N=42) | Unlabeled TST (N=36) | Unlabeled TST Crossover (N=19)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0 | 4
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 2
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant mesenteric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 2 | 1 | 0
Sepsis (Infections and infestations) | 1 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1
Cystitis (Infections and infestations) | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0
Endocarditis bacterial (Infections and infestations) | 0 | 1 | 0
Fungaemia (Infections and infestations) | 0 | 1 | 0
Proteus infection (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypothermia (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Ulcer (General disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TST and Iodine I 131 TST (N=42) | Unlabeled TST (N=36) | Unlabeled TST Crossover (N=19)
Fatigue (General disorders) | 16 | 12 | 8
Pyrexia (General disorders) | 11 | 7 | 3
Chills (General disorders) | 10 | 7 | 3
Malaise (General disorders) | 4 | 1 | 1
Pain (General disorders) | 2 | 3 | 1
Feeling hot (General disorders) | 3 | 2 | 0
Oedema peripheral (General disorders) | 2 | 2 | 1
Asthenia (General disorders) | 2 | 2 | 0
Chest pain (General disorders) | 3 | 1 | 0
Chest discomfort (General disorders) | 2 | 1 | 0
Discomfort (General disorders) | 1 | 1 | 1
Influenza like illness (General disorders) | 1 | 1 | 1
Facial pain (General disorders) | 0 | 2 | 0
Local swelling (General disorders) | 1 | 1 | 0
Application site erythema (General disorders) | 1 | 0 | 0
Axillary pain (General disorders) | 1 | 0 | 0
Catheter site related reaction (General disorders) | 1 | 0 | 0
Fat tissue increased (General disorders) | 0 | 1 | 0
Gait disturbance (General disorders) | 1 | 0 | 0
Infusion site extravasation (General disorders) | 1 | 0 | 0
Infusion site reaction (General disorders) | 1 | 0 | 0
Infusion site swelling (General disorders) | 1 | 0 | 0
Injection site extravasation (General disorders) | 0 | 1 | 0
Nodule (General disorders) | 1 | 0 | 0
Oedema (General disorders) | 1 | 0 | 0
Secretion discharge (General disorders) | 1 | 0 | 0
Swelling (General disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 21 | 6 | 2
Diarrhoea (Gastrointestinal disorders) | 6 | 3 | 1
Abdominal discomfort (Gastrointestinal disorders) | 3 | 2 | 2
Constipation (Gastrointestinal disorders) | 2 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 4 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 1
Flatulence (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 1 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 1 | 0
Retching (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 6 | 2 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 3 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 2 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 3 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Ingrown skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 2 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 2
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
WBC <2000 cells/mm^3 (Investigations) | 18 | 4 | 11
ANC <1000 cells/mm^3 (Investigations) | 14 | 4 | 11
Platelets <50000 cells/mm^3 (Investigations) | 15 | 1 | 9
Hemoglobin <8.0 g/dL (Investigations) | 6 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 7 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 6 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 4 | 1
Bronchitis (Infections and infestations) | 1 | 3 | 1
Pneumonia (Infections and infestations) | 1 | 2 | 0
Herpes simplex (Infections and infestations) | 1 | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 1 | 1
Folliculitis (Infections and infestations) | 1 | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 2
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0
Fungal skin infection (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0
Urinary tract infection enterococcal (Infections and infestations) | 1 | 0 | 0
Varicella (Infections and infestations) | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Gingival infection (Infections and infestations) | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 1
Headache (Nervous system disorders) | 5 | 7 | 4
Dizziness (Nervous system disorders) | 3 | 3 | 0
Paraesthesia (Nervous system disorders) | 1 | 1 | 1
Somnolence (Nervous system disorders) | 1 | 1 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0
Burning sensation (Nervous system disorders) | 0 | 1 | 0
Dizziness postural (Nervous system disorders) | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 0 | 0
Mental impairment (Nervous system disorders) | 1 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 6 | 0 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 0 | 3
Lymphadenopathy (Blood and lymphatic system disorders) | 3 | 4 | 0
Lymph node pain (Blood and lymphatic system disorders) | 2 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 2 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Body temperature increased (Investigations) | 3 | 1 | 0
Weight decreased (Investigations) | 2 | 0 | 2
Cardiac murmur (Investigations) | 1 | 1 | 0
Bacterial test positive (Investigations) | 0 | 1 | 0
Blood potassium decreased (Investigations) | 0 | 1 | 0
Breath sounds abnormal (Investigations) | 1 | 0 | 0
Heart rate increased (Investigations) | 1 | 0 | 0
Red blood cell count decreased (Investigations) | 1 | 0 | 0
Transaminases increased (Investigations) | 1 | 0 | 0
Weight increased (Investigations) | 1 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 4 | 3 | 1
Anxiety (Psychiatric disorders) | 2 | 1 | 1
Depression (Psychiatric disorders) | 0 | 2 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 6 | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Flushing (Vascular disorders) | 2 | 1 | 0
Hypotension (Vascular disorders) | 1 | 1 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 3 | 0 | 0
Atrial tachycardia (Cardiac disorders) | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 3 | 0 | 3
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 2
Dysuria (Renal and urinary disorders) | 1 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 0 | 1 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 1
Nocturia (Renal and urinary disorders) | 0 | 0 | 1
Ear pruritus (Ear and labyrinth disorders) | 1 | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 1
Dry eye (Eye disorders) | 1 | 0 | 0
Eye irritation (Eye disorders) | 1 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 1 | 0
Ocular icterus (Eye disorders) | 1 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Nipple pain (Reproductive system and breast disorders) | 1 | 0 | 0
Prostatism (Reproductive system and breast disorders) | 0 | 1 | 0
Graft versus host disease (Immune system disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.